CLINICAL TRIAL: NCT01334502
Title: A Phase I and Feasibility Study of Everolimus (RAD001) Plus R-CHOP for New Untreated Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Everolimus, Rituximab, and Combination Chemotherapy in Treating Patients With Newly Diagnosed Untreated Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N1085; NCCTG-N1085; CDR0000698584 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-02643 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Everolimus; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- everolimus and RCHOP (Experimental): Patients registered to the study will receive an assigned dose of everolimus by mouth and RCHOP for a maximum of six cycles. Each cycle is a total of 21 days. RCHOP consists of 375 mg/m2 IV rituximab, 750 mg/m2 IV cyclophosphamide, 50 mg/m2 IV doxorubicin, 1.4 mg/m2 IV vincristine and 100 mg/m2 by mouth QD prednisone. The study includes a Phase I component to determine the maximum tolerated dose of everolimus and the second component determines the feasibility of therapy administered to lymphoma patients.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: everolimus; Drug: prednisone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: rituximab — PO
Drug: cyclophosphamide — IV
Drug: doxorubicin hydrochloride — IV
Drug: everolimus — PO
Drug: prednisone — PO
Drug: vincristine sulfate — IV

SUMMARY:
RATIONALE: Everolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, can block cancer cells in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or stopping them from dividing. Giving everolimus together with rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and the best dose of everolimus when given together with rituximab and combination chemotherapy in treating patients with newly diagnosed untreated diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish the maximum-tolerated dose (MTD) of everolimus in combination with R-CHOP (rituximab, cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate and prednisone) chemotherapy.
* To assess the feasibility of everolimus in combination with standard R-CHOP chemotherapy in patients with newly diagnosed diffuse large B-cell lymphoma.

Secondary

* To describe the toxicities associated with everolimus in combination with R-CHOP chemotherapy.
* To further describe the toxicities associated with everolimus in combination with R-CHOP chemotherapy.
* To assess the rate of event-free survival (EFS) at 12 months for diffuse large B-cell lymphoma patients treated with everolimus in combination with R-CHOP chemotherapy.
* To evaluate overall response rate, complete response rate, duration of response, EFS, overall survival, and progression-free survival for patients treated with everolimus in combination with R-CHOP chemotherapy.

Tertiary

* To profile gene expression using immunohistochemistry and categorize patients as germinal-center B-cell-like (GBC) vs activated B-cell-like (ABC) vs unclassified lymphoma subtype. (exploratory)
* To determine whether previously identified predictive markers in large cell lymphoma remain valid with the addition of everolimus to R-CHOP chemotherapy. (exploratory)

OUTLINE: This is a multicenter, dose-escalation study of everolimus followed by a feasability expanded-cohort study.

Patients receive everolimus orally (PO) once daily (QD) on days 1-10 or 1-14; rituximab IV, cyclophosphamide IV, doxorubicin hydrochloride IV over 15-60 minutes, and vincristine sulfate IV on day 1; and prednisone PO QD on days 1-5. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Tumor biopsies are collected for laboratory studies and patients may undergo blood and needle biopsy sample collection for correlative studies.

After completion of study treatment, patients are followed up every 3-6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Untreated, histological diagnosis of CD20-positive diffuse large B-cell lymphoma
* Stage II-IV (Ann Arbor Staging)
* Measurable or assessable disease defined as at least one of the following:

  * A lymph node or tumor mass that is ≥ 2.0 cm in at least one dimension by CT portion of PET/CT scan, CT scan, or MRI
  * Diffuse infiltration of an organ such as the stomach, bone marrow, peripheral blood, liver, lungs, or bowel by lymphoma without a discrete mass would constitute assessable, but not measurable, disease
* Diagnostic tissue slides and paraffin-embedded block must be available
* No CNS lymphoma or cerebrospinal fluid involvement with malignant lymphoma cells

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1,500/mm³
* Peripheral platelet count ≥ 100,000/mm³
* Hemoglobin (HgB) > 9.0 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)

  * For total bilirubin > 1.5 times ULN, the direct bilirubin must be normal
* Alkaline phosphatase ≤ 3 times ULN (≤ 5 times ULN if evidence of direct liver involvement by lymphoma)
* AST ≤ 3 times ULN (≤ 5 times ULN if evidence of direct liver involvement by lymphoma)
* Creatinine ≤ ULN
* Negative serum or urine pregnancy test
* Not pregnant or nursing
* Men or women of childbearing potential must be willing to employ adequate contraception throughout the study and for12 months after the last dose of study drug
* Willing to return to the National Central Cancer Treatment Group (NCCTG) enrolling institution for follow-up
* Willing to provide archival tissue from the primary diagnosis (original lymphoma lymph node tissue biopsy)
* Willing to abstain from eating grapefruit or drinking grapefruit juice for the duration of the study
* Diabetic patients who are taking insulin or oral anti-diabetic therapy must have HbA1c ≤ 8%, or a fasting serum glucose ≤ 110% ULN
* HIV-positive patients must have CD4 count ≥ 400/mm³
* No co-morbid systemic illnesses or other severe concurrent disease that, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* No immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be HIV positive with a CD4 count of < 400/mm³
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Severely impaired lung function
  * Uncontrolled diabetes as defined by fasting serum glucose > 1.5 times ULN

    * Optimal glycemic control should be achieved before starting trial therapy
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Liver disease such as cirrhosis or severe hepatic impairment
  * Chronic active hepatitis
  * Chronic persistent hepatitis or history of hepatitis B or C
* No other active malignancy except non-melanotic skin cancer or carcinoma in situ of the cervix

  * If there is a history of prior malignancy, patients must not be receiving other specific treatment (other than hormonal therapy) for their cancer
* No positive hepatitis B antigen (HBsAg) or hepatitis C serology (HCV) tests meeting the following criteria:

  * Hepatitis B surface antigen (HbsAg) and antibody to hepatitis B core (anti-HBc) or hepatitis C antibody
  * All patients must be screened prior to registration
  * Patients who have evidence of chronic or acute infection with either hepatitis B or C may not be treated on this protocol

PRIOR CONCURRENT THERAPY:

* Not receiving any other investigational agent that would be considered as a treatment for the primary neoplasm
* No planned immunization with attenuated live vaccines ≤ 7 days prior to registration or during study period

  * Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus
  * Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella, and TY21a typhoid vaccines
* Not currently on enzyme-inducing anti-convulsants or other strong inducers of CYP3A4 (efavirenz, nevirapine, barbiturates, carbamazepine, modafinil, phenobarbital, phenytoin, rifabutin, rifampin, pioglitazone, or St. John wort) or strong inhibitors of CYP3A4 (indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, saquinavir, or telithromycin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
MTD of everolimus in combination with R-CHOP | Up to 15 months post registration to Phase I portion of the study
Adverse events profile | Up to 15 months post registration to Phase I portion of the study
Toxicity profile | Up to 15 months post registration to Phase I portion of the study
Proportion of patients who have a significant toxicity | Up to 2.5 years post registration to Feasibility portion of the study

SECONDARY OUTCOMES:
Rate of EFS | Up to 5 years post treatment of the feasibility portion of the study
Overall response rate, CR rate, overall survival, PFS, and duration of response | Up to 5 years post treatment of the feasibility portion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Johnston, MD, PhD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic Cancer Center, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Johnston PB, LaPlant B, McPhail E, Habermann TM, Inwards DJ, Micallef IN, Colgan JP, Nowakowski GS, Ansell SM, Witzig TE. Everolimus combined with R-CHOP-21 for new, untreated, diffuse large B-cell lymphoma (NCCTG 1085 [Alliance]): safety and efficacy results of a phase 1 and feasibility trial. Lancet Haematol. 2016 Jul;3(7):e309-16. doi: 10.1016/S2352-3026(16)30040-0. Epub 2016 Jun 5. PMID 27374464